CLINICAL TRIAL: NCT06861179
Title: Basic and Clinical Studies on the Effects of the Formulation of Compound Phellinus Igniarius Decoction on Radiation Pneumonitis
Brief Title: The Formulation of Compound Phellinus Igniarius Decoction on Radiation Pneumonitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Feng Wei, Director, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022QJF0101
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Radiation Pneumonitis
MeSH Terms: conditions — Radiation Pneumonitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the effects of The formulation of Compound Phellinus igniarius decoction on radiation pneumonitis (Experimental): The patients were randomly allocated into two groups, each comprising 20 patients. All patients received with DT: 50-60 Gy/20-30F thoracic radiotherapy, all with 6mv linear accelerator irradiation. The study group was defined as receiving the formulation of Compound Phellinus igniarius decoction, 150ml bid was administered continuously until the end of radiotherapy.
  Interventions: Drug: The formulation of Compound Phellinus igniarius decoction
- The formulation of Compound Phellinus igniarius decoction on radiation pneumonitis (No Intervention): he patients were randomly allocated into two groups, each comprising 20 patients. All patients received with DT: 50-60 Gy/20-30F thoracic radiotherapy, all with 6mv linear accelerator irradiation. The control group was defined as receiving standard-dose radiotherapy without the administration of the formulation of Compound Phellinus igniarius decoction.

INTERVENTIONS:
Drug: The formulation of Compound Phellinus igniarius decoction — The formulation of Compound Phellinus igniarius decoction is manufactured by Hangzhou Qianjifang Technology Co., Ltd, the composition includes Phellinus igniarius 12g, jujube 3g, wolfberry 3g, tangerine peel 1g. The dosage regimen was as follows: 4 Packs of the formulation of Compound Phellinus igniarius decoction (Phellinus igniarius Herbal Decoction Pieces) + 1 Pack of the formulation of Compound Phellinus igniarius decoction(Excipients) per day, administered twice daily throughout the entire course of radiotherapy until its completion.
  Arms: the effects of The formulation of Compound Phellinus igniarius decoction on radiation pneumonitis

SUMMARY:
The objectives of this clinical trial were to determine the radioprotective effects and underlying biological mechanisms of Phellinus igniarius and its active components during radiotherapy in patients with thoracic malignant tumors.

The study group was given the formulation of Compound Phellinus igniarius decoction daily during radiotherapy, 150ml bid until the end of radiotherapy; The control group only received standard dose radiotherapy without the formulation of Compound Phellinus igniarius decoction intervention.

The baseline differences between the two groups were compared, including gender, smoking history, body mass index (BMI), pathological classification, median age of onset, inflammatory factors, tumor markers, TNM stage, KPS score, fatigue score, incidence and grade of radiation pneumonitis, incidence of other radiotherapy-related adverse reactions, and average radiation dose.

DETAILED DESCRIPTION:
Investigators measured the levels of inflammatory factors and tumor markers in blood samples of patients in the two income groups, and administered questionnaires on the degree of fatigue and general status of patients. Metabolite changes and gut microbiota homeostasis in patient fecal samples were then detected by untargeted metabolomics and metagenomics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, ECOG score≤2, possess adequate communication and comprehension abilities, and have an anticipated survival time exceeding 6 months
* Confirmed diagnosis of lung malignancy through imaging and pathological examination
* Indications for thoracic radiotherapy, DT:50-60Gy/20-30F
* Normal function of vital organs, including the heart, liver, kidneys, and gastrointestinal system

Exclusion Criteria:

* Patients with pre-existing pulmonary conditions, including idiopathic pulmonary fibrosis
* Individuals with systemic immune disorders
* Those with concurrent major infections
* Patients diagnosed with hematological disorders. All participants provided written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Inflammatory factors in blood samples of patients in the study group | Blood samples were collected from patients 1-3 days before the start of RT and one month after the end of RT
  The Concentration of IL-1β、IL-6、IL-8、IL-2、IL-4、IL-5
Tumor markers in blood samples of patients in the study group | Blood samples were collected from patients 1-3 days before the start of RT, and one month after the end of RT
  The Levels of NSE、CYFRA21-1、SCCA、CA-125、CA-199、CEA

CONTACTS AND LOCATIONS:
Overall Officials: Wei Feng, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen H, Tian T, Miao H, Zhao YY. Traditional uses, fermentation, phytochemistry and pharmacology of Phellinus linteus: A review. Fitoterapia. 2016 Sep;113:6-26. doi: 10.1016/j.fitote.2016.06.009. Epub 2016 Jun 23. PMID 27343366
- [Background] Ni Z, Li J, Qian X, Yong Y, Wu M, Wang Y, Lv W, Zhang S, Zhang Y, Shao Y, Chen A. Phellinus igniarius Polysaccharides Ameliorate Hyperglycemia by Modulating the Composition of the Gut Microbiota and Their Metabolites in Diabetic Mice. Molecules. 2023 Oct 17;28(20):7136. doi: 10.3390/molecules28207136. PMID 37894615
- [Background] Zhong S, Sun YQ, Huo JX, Xu WY, Yang YN, Yang JB, Wu WJ, Liu YX, Wu CM, Li YG. The gut microbiota-aromatic hydrocarbon receptor (AhR) axis mediates the anticolitic effect of polyphenol-rich extracts from Sanghuangporus. Imeta. 2024 Mar 11;3(2):e180. doi: 10.1002/imt2.180. eCollection 2024 Apr. PMID 38882491